CLINICAL TRIAL: NCT04620798
Title: Longitudinal COVID-19 Antibody Testing in Indiana University Undergraduate Students
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indiana University (Other)
Responsible Party: Principal Investigator, Molly Rosenberg, Assistant Professor Public Health, Indiana University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: 2008293852
Record Dates: First submitted 2020-11-04; First posted 2020-11-09 (Actual); Results first posted 2022-01-31 (Actual); Last update posted 2022-01-31 (Actual); Status verified 2022-01

CONDITIONS: SARS-CoV-2; Serology; Students

STUDY DESIGN:
Intervention Model Description: Participants will be randomized to receive their antibody test results either within a day of the test or after a four-week waiting period in order to assess whether receiving the results of an antibody test changes protective behavior to avoid SARS-CoV-2 infections.
Who Masked: Participant, Investigator
Masking Description: Because we are attempting to assess the impact of having knowledge about a participants' antibody test result on their engagement in protective behaviors to avoid SARS-CoV-2 infections, the intervention information will be masked from the participant and the investigators.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will be given their results of their antibody test immediately (within 24 hours) and will be followed and surveyed to see if having this knowledge changes their engagement with SARS-CoV-2 prevention behaviors.
  Interventions: Behavioral: Immediate vs. delayed provision of antibody test results
- Control (Delayed) (No Intervention): Participants will be given their results of their antibody test after 4 weeks. Their engagement with SARS-CoV-2 prevention behaviors will also be assessed following testing.

INTERVENTIONS:
Behavioral: Immediate vs. delayed provision of antibody test results — The primary experiment will be assessing whether provision of the antibody test results leads to behavior change with respect to personal protective behaviors. To that end, we will randomize all participants to a trial arm that immediately receive results (within 24 hours) or a trial arm with a delayed provision of results (after 4 weeks).
  Arms: Intervention

SUMMARY:
The primary goal for this study is to assess whether receiving the results of an antibody test changes protective behavior to avoid SARS-CoV-2 infections (i.e., mask-wearing, physical distancing, limiting close contacts/avoiding crowds, hand-washing, avoiding contact with high-risk individuals). While studies have been published on the cross-sectional relationship between risk perception and other demographic characteristics and health behaviors that are protective for SARS-CoV-2 infection (see citations), there have been no studies showing the effect of receiving information about antibody positivity on protective behavior. Not only can results from this study be used to better model transmission, a better understanding of college student's risk perception around SARS-CoV-2 infections has implications for future vaccination strategies as well. There are concerns that a desire to return to "normal" life in combination with reduced perception of risk could have negative consequences for uptake of vaccination (Johns Hopkins Center for Health Security 2020 report, The Public's Role in COVID-19 Vaccination: Planning Recommendations Informed by Design Thinking and the Social, Behavioral, and Communication Sciences).

The antibody test used in this study is named 'SARS-CoV-2 IgM/IgG rapid assay kit (Colloidal Gold)'. It provides a fast, on-site, and accurate detection of IgM/IgG antibodies against SARS-CoV-2, with positive results of IgM antibodies indicating a recent infection, while positive results of IgG antibodies signaling a longer or previous infection. It can detect IgM and IgG antibodies against SARS-CoV-2 in human specimens of serum, plasma, or venous whole blood.

DETAILED DESCRIPTION:
This study will take place between September - November, 2020, and will ask participants to participate in: a web-based baseline survey, two rounds of SARS-CoV-2 serological testing (September and November), and bi-weekly web-based behavioral surveys (4 total surveys). Each is described in more detail below:

Web-based baseline survey: The baseline survey is designed to collect data on participant demographics, SARS-CoV-2 protective behaviors, alcohol drinking habits, nicotine use, and personality profile and should take less than 30 minutes to fill out. Participants who provide informed consent will be provided the link to the survey which they can fill out at a time convenient to them prior to first round of serological testing.

SARS-CoV-2 serological testing: There will be two rounds of SARS-CoV-2 serological testing, once at baseline (September 14-23) and once at endline (November 9-11). The serological testing visits will involve in-person laboratory testing for SARS-CoV-2 antibodies. The laboratory test involves a fingerstick to provide a small blood sample for the antibody test kits.

Antibody test results will eventually be provided to all study participants via secure link sent by email. With this message, we will include a clearly written information sheet about the chance for inaccurate test results and how it is still unknown whether previous infections confer immunity to future infections. We will clearly counsel participants to not use the results of the tests as proof of a previous SARS-CoV-2 infection, nor as a reason to change their behaviors. If participants wish to participate in the study, but do not wish to be provided with their antibody test results, they will be able to opt out of the results provision. If any participants opt out of receiving their test results, these participants would essentially create a third category of respondents: those who do not receive their results at all. However, these participants will still be analyzed with the trial arm to which they were randomized (intent to treat analysis).

The primary experiment will assess whether provision of the antibody test results leads to behavior change with respect to personal protective behaviors. To that end, all participants will be randomized to a trial arm that immediately receive results (within 24 hours) or a trial arm with a delayed provision of results (after 4 weeks). So as to not incentivize early drop-out, if a participant in the delayed results arm drops out early, they will still be provided their test results at the regularly scheduled time, not earlier. All other procedures between arms are identical. The endline laboratory test results will be delivered to all participants in the same timeframe - within 24-72 hours. The early and delayed test result intervention will have completed after the first round of testing.

Web-based behavioral surveys: To assess whether or not the provision of antibody test results changes behaviors, participants will self-reported behaviors in a short web-based survey every two weeks under observation. Links to these surveys will be sent to participants at regular bi-weekly intervals. Participants will fill out these short follow-up surveys on their computers or mobile devices. They are designed to take about 5 minutes or less to complete for each survey.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older
* Current IU undergraduate student
* Current resident of Monroe County, Indiana

Exclusion Criteria:

* Younger than 18 years old
* Current residence outside of Monroe County, Indiana

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1076 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2020-11-11 (Actual); Study Completion 2020-11-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Molly Rosenberg, PhD, Principal Investigator — Indiana University Department of Epidemiology and Biostatistics
Locations (1):
- Indiana University, Bloomington, Indiana, United States

IPD SHARING:
Plan to Share IPD: Yes
The study team will make the following documents available to the public upon completion of the study: (1) Study Protocol, (2) Statistical Analysis Plan (SAP), (3) Informed Consent Form (ICF), and (4) Clinical Study Report (CSR). The individual participant data as well as the analytic code will not be made available to the public due to privacy concerns and in order to protect participants' private health information but will be available from the Principal Investigator upon request.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: These study protocol documents will be made available upon completion of the study and the analyses. A de-identified, limited data set and analytic code will be available from the Principal Investigator upon request.
Access Criteria: Protocol will be available on clinicaltrials.gov while the other documents, data, and analytic code from the Principal Investigator upon request.

REFERENCES:
- [Derived] Chen C, Rosenberg M, Li M, Macy JT, Ludema C. Patterns and persistence of SARS-CoV-2 seropositivity among college students at Indiana University-Bloomington. BMJ Open. 2025 Sep 22;15(9):e091418. doi: 10.1136/bmjopen-2024-091418. PMID 40983579
- [Derived] Kianersi S, Luetke M, Ludema C, Valenzuela A, Rosenberg M. Use of research electronic data capture (REDCap) in a COVID-19 randomized controlled trial: a practical example. BMC Med Res Methodol. 2021 Aug 21;21(1):175. doi: 10.1186/s12874-021-01362-2. PMID 34418958

RESULTS

PARTICIPANT FLOW:
Recruitment Details: We randomly sampled 7,499 students from the sampling frame of all IU Bloomington undergraduates enrolled at the beginning of the Fall 2020 semester. Students in the sample were eligible to participate if they were (1) aged 18 years or older, (2) a current IU Bloomington undergraduate student, and (3) currently residing in Monroe County, Indiana. Of those sampled, 4,069 potential participants met the inclusion criteria for the study and were contacted by email with a study invitation.
Pre-assignment Details: Following the study invitation, 1076 of the 4069 eligible sampled students were enrolled in the study and received randomization. 2651 students tacitly refused participation, 21 students explicitly refused participation or withdrew from the study, and 321 students missed the baseline study visit.
Groups:
- Intervention (Immediate Results): Participants will be given their results of their antibody test immediately (within 24 hours).
- Control (Delayed Results): Participants will be given their results of their antibody test four weeks following the test.
Period: Overall Study
Arm/Group | Intervention (Immediate Results) | Control (Delayed Results)
Started (Includes all eligible participants who consented to enrollment and were randomized to received either immediate or delayed results.) | 536 | 540
Completed Behavioral Survey (Includes all participants who completed the behavioral survey two weeks following baseline antibody testing.) | 477 | 508
Completed (Includes all participants who completed endline antibody testing eight weeks following baseline antibody testing.) | 410 | 402
Not Completed | 126 | 138
Not completed — Lost to Follow-up | 126 | 138

BASELINE CHARACTERISTICS:
Population: Indiana University Bloomington undergraduate students enrolled at the beginning of the Fall 2020 semester.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention (Immediate Results) | Control (Delayed Results) | Total
Number analyzed (Participants) | 536 | 540 | 1076
Age, Categorical [Count of Participants; unit: Participants] — Population: Only includes participants who self-reported their age at baseline (66 participants were missing this data).
  Participants
    number analyzed (Participants) | 508 | 502 | 1010
    <=18 years | 0 | 0 | 0
    Between 18 and 65 years | 508 | 502 | 1010
    >=65 years | 0 | 0 | 0
Age, Customized [Count of Participants; unit: Participants]
  Age, Categorical: 18 years old | 111 | 97 | 208
  Age, Categorical: 19 years old | 109 | 115 | 224
  Age, Categorical: 20 years old | 109 | 119 | 228
  Age, Categorical: 21 years old | 132 | 123 | 255
  Age, Categorical: 22+ years old | 47 | 48 | 95
  Age, Categorical: Missing | 28 | 38 | 66
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Only includes participants who self-reported information regarding their biological sex at birth (five participants were missing this data).
  Participants
    number analyzed (Participants) | 534 | 537 | 1071
    Female | 333 | 356 | 689
    Male | 201 | 181 | 382
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 39 | 39 | 78
  Not Hispanic or Latino | 497 | 501 | 998
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 43 | 37 | 80
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 6 | 7 | 13
  White | 417 | 430 | 847
  More than one race | 43 | 42 | 85
  Unknown or Not Reported | 27 | 24 | 51
Region of Enrollment [Number; unit: participants]
  United States | 536 | 540 | 1076
Undergraduate School Year [Count of Participants; unit: Participants] — Participant year of enrollment in school as of Fall 2020.
  Participants
    First Year | 123 | 113 | 236
    Second Year | 119 | 127 | 246
    Third Year | 127 | 137 | 264
    Fourth Year | 154 | 143 | 297
    Fifth Year or More | 10 | 17 | 27
    Missing | 3 | 3 | 6
Residence [Count of Participants; unit: Participants] — Participant lives in on-campus or off-campus housing.
  Participants
    On-Campus | 176 | 162 | 338
    Off-Campus | 358 | 375 | 733
    Missing | 2 | 3 | 5
Greek Affiliation Status [Count of Participants; unit: Participants] — Participant actively participates in campus Greek life (i.e., is a member of a sorority or fraternity).
  Participants
    Yes | 129 | 129 | 258
    No | 403 | 409 | 812
    Missing | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Frequency of Handwashing
Description: This outcome was dichotomized into Always and Very Often versus Sometimes, Rarely, and Never. It will be self-reported in a web-based follow-up survey administered at 2 weeks after the baseline antibody test, with an item adapted from the WHO 2020 "Monitoring knowledge, risk perceptions, preventive behaviours and trust to inform pandemic outbreak response":
  "During the last 7 days, which of the following measures have you taken to prevent infection from COVID-19?"
  -Frequently washed my hands with soap and water for at least 20 seconds
  Response options are: Always, Very Often, Sometimes, Rarely, Never
Time Frame: 2 weeks after the baseline antibody test
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (Immediate Results) | Control (Delayed Results)
Number analyzed (Participants) | 477 | 508
Participants
  Always or Very Often | 412 | 432
  Never, Sometimes, or Rarely | 65 | 75
  Not Applicable | 0 | 1
Statistical Analysis 1: Comparison: Intervention (Immediate Results) vs Control (Delayed Results); This analysis includes only those participants with a negative antibody test result at baseline to test the association between the treatment condition (immediate vs. delayed test results) and behavioral outcomes. The reference group for this analysis was the control (delayed results) group; Test type: Superiority; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.96 to 1.07] — This analysis compares the probability of responding "Very Often/Always" vs. all other response categories. The reference group for this analysis was the control (delayed results) group
Statistical Analysis 2: Comparison: Intervention (Immediate Results) vs Control (Delayed Results); This analysis uses only those participants with a positive antibody test result at baseline to test the association between the treatment condition (immediate vs. delayed test results) and behavioral outcomes. The reference group for this analysis was the control (delayed results) group; Test type: Superiority; Risk Ratio (RR) = 1.05, 95% CI 2-sided [0.77 to 1.44] — [estimate comment as in outcome 1, analysis 1]

2. Primary Outcome: Frequency of Face Touching
Description: This outcome was dichotomized into Always and Very Often versus Sometimes, Rarely, and Never. This outcome will be self-reported in a web-based follow-up survey administered at 2 weeks after the baseline antibody test, with an item adapted from the WHO 2020 "Monitoring knowledge, risk perceptions, preventive behaviours and trust to inform pandemic outbreak response":
  "During the last 7 days, which of the following measures have you taken to prevent infection from COVID-19?"
  -Avoided touching my eyes, nose and mouth with unwashed hands
  Response options are: Always, Very Often, Sometimes, Rarely, Never
Time Frame: 2 weeks after the baseline antibody test
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (Immediate Results) | Control (Delayed Results)
Number analyzed (Participants) | 476 | 507
Participants
  Always or Very Often | 280 | 303
  Never, Sometimes, or Rarely | 196 | 204
Statistical Analysis 1: Comparison: Intervention (Immediate Results) vs Control (Delayed Results); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 0.99, 95% CI 2-sided [0.89 to 1.10] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Intervention (Immediate Results) vs Control (Delayed Results); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 0.90, 95% CI 2-sided [0.50 to 1.62] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: Frequency of Hand Sanitizer Use
Description: This outcome was dichotomized into Always and Very Often versus Sometimes, Rarely, and Never. This outcome will be self-reported in a web-based follow-up survey administered at 2 weeks after the baseline antibody test, with an item adapted from the WHO 2020 "Monitoring knowledge, risk perceptions, preventive behaviours and trust to inform pandemic outbreak response":
  "During the last 7 days, which of the following measures have you taken to prevent infection from COVID-19?"
  -Used disinfectants or hand sanitizer to clean hands when soap and water were not available
  Response options are: Always, Very Often, Sometimes, Rarely, Never
Time Frame: 2 weeks after the baseline antibody test
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (Immediate Results) | Control (Delayed Results)
Number analyzed (Participants) | 477 | 505
Participants
  Always or Very Often | 414 | 436
  Never, Sometimes, or Rarely | 60 | 69
  Not Applicable | 3 | 0
Statistical Analysis 1: Comparison: Intervention (Immediate Results) vs Control (Delayed Results); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.96 to 1.06] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Intervention (Immediate Results) vs Control (Delayed Results); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 0.98, 95% CI 2-sided [0.74 to 1.31] — [estimate comment as in outcome 1, analysis 1]

4. Primary Outcome: Frequency of Social Event Avoidance
Description: This outcome was dichotomized into Always and Very Often versus Sometimes, Rarely, and Never. It will be self-reported in a web-based follow-up survey administered at 2 weeks after the baseline antibody test, with an item adapted from the WHO 2020 "Monitoring knowledge, risk perceptions, preventive behaviours and trust to inform pandemic outbreak response":
  "During the last 7 days, which of the following measures have you taken to prevent infection from COVID-19?"
  -Avoided a social event I wanted to attend
  Response options are: Always, Very Often, Sometimes, Rarely, Never
Time Frame: 2 weeks after the baseline antibody test
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (Immediate Results) | Control (Delayed Results)
Number analyzed (Participants) | 477 | 507
Participants
  Always or Very Often | 209 | 236
  Never, Rarely, or Sometimes | 224 | 228
  Not Applicable | 44 | 43
Statistical Analysis 1: Comparison: Intervention (Immediate Results) vs Control (Delayed Results); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 0.96, 95% CI 2-sided [0.84 to 1.09] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Intervention (Immediate Results) vs Control (Delayed Results); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 0.75, 95% CI 2-sided [0.33 to 1.72] — This analysis compares the probability of a response of "Very Often/Always" vs. all other response categories. The reference group for this analysis was the control (delayed results) group

5. Primary Outcome: Frequency of Staying Home From Work/School
Description: This outcome is dichotomized into Always and Very Often versus Sometimes, Rarely, and Never. It will be self-reported in a web-based follow-up survey administered at 2 weeks after the baseline antibody test, with an item adapted from the WHO 2020 "Monitoring knowledge, risk perceptions, preventive behaviours and trust to inform pandemic outbreak response":
  "During the last 7 days, which of the following measures have you taken to prevent infection from COVID-19?"
  -Stayed at home from work/school
  Response options are: Always, Very Often, Sometimes, Rarely, Never
Time Frame: 2 weeks after the baseline antibody test
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (Immediate Results) | Control (Delayed Results)
Number analyzed (Participants) | 477 | 506
Participants
  Always or Very Often | 152 | 185
  Never, Rarely, or Sometimes | 254 | 255
  Not Applicable | 71 | 66
Statistical Analysis 1: Comparison: Intervention (Immediate Results) vs Control (Delayed Results); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 0.87, 95% CI 2-sided [0.74 to 1.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Intervention (Immediate Results) vs Control (Delayed Results); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 1.40, 95% CI 2-sided [0.60 to 3.25] — [estimate comment as in outcome 4, analysis 2]

6. Primary Outcome: Frequency of Mask Wearing
Description: This outcome is dichotomized into Always versus Very Often, Sometimes, Rarely, and Never. It will be self-reported in a web-based follow-up survey administered at 2 weeks after the baseline antibody test, with an item adapted from the WHO 2020 "Monitoring knowledge, risk perceptions, preventive behaviours and trust to inform pandemic outbreak response":
  "During the last 7 days, which of the following measures have you taken to prevent infection from COVID-19?"
  -Wore a mask in public
  Response options are: Always, Very Often, Sometimes, Rarely, Never
Time Frame: 2 weeks after the baseline antibody test
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (Immediate Results) | Control (Delayed Results)
Number analyzed (Participants) | 476 | 504
Participants
  Always | 400 | 433
  Never, Rarely, Sometimes, or Very Often | 76 | 71
Statistical Analysis 1: Comparison: Intervention (Immediate Results) vs Control (Delayed Results); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.99 to 1.03] — This analysis compares the probability of a response of "Always" vs. all other response categories. The reference group for this analysis was the control (delayed results) group
Statistical Analysis 2: Comparison: Intervention (Immediate Results) vs Control (Delayed Results); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 0.97, 95% CI 2-sided [0.77 to 1.21] — [estimate comment as in outcome 6, analysis 1]

7. Primary Outcome: Frequency of Physical Distancing
Description: This outcome is dichotomized into Always and Very Often versus Sometimes, Rarely, and Never. It will be self-reported in a web-based follow-up survey administered at 2 weeks after the baseline antibody test, with an item adapted from the WHO 2020 "Monitoring knowledge, risk perceptions, preventive behaviours and trust to inform pandemic outbreak response":
  "During the last 7 days, which of the following measures have you taken to prevent infection from COVID-19?"
  -Ensured physical distancing in public
  Response options are: Always, Very Often, Sometimes, Rarely, Never
Time Frame: 2 weeks after the baseline antibody test
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (Immediate Results) | Control (Delayed Results)
Number analyzed (Participants) | 477 | 506
Participants
  Always or Very Often | 427 | 452
  Never, Rarely, or Sometimes | 50 | 54
Statistical Analysis 1: Comparison: Intervention (Immediate Results) vs Control (Delayed Results); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 1.01, 95% CI 2-sided [0.97 to 1.06] — [estimate comment as in outcome 4, analysis 2]
Statistical Analysis 2: Comparison: Intervention (Immediate Results) vs Control (Delayed Results); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 0.82, 95% CI 2-sided [0.60 to 1.11] — [estimate comment as in outcome 4, analysis 2]

8. Primary Outcome: Frequency of Avoiding People at High-risk for Severe COVID-19 Infections
Description: This outcome was dichotomized into Always and Very Often versus Sometimes, Rarely, and Never. This outcome will be self-reported in a web-based follow-up survey administered at 2 weeks after the baseline antibody test, with an item adapted from the WHO 2020 "Monitoring knowledge, risk perceptions, preventive behaviours and trust to inform pandemic outbreak response":
  "During the last 7 days, which of the following measures have you taken to prevent infection from COVID-19?"
  -Avoided contact with people at high-risk for severe COVID-19 infections
  Response options are: Always, Very Often, Sometimes, Rarely, Never
Time Frame: 2 weeks after the baseline antibody test
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (Immediate Results) | Control (Delayed Results)
Number analyzed (Participants) | 477 | 507
Participants
  Always or Very Often | 433 | 466
  Never, Sometimes, or Rarely | 30 | 31
  Not Applicable | 14 | 10
Statistical Analysis 1: Comparison: Intervention (Immediate Results) vs Control (Delayed Results); [analysis description as in outcome 1, analysis 1]; Test type: Superiority; Risk Ratio (RR) = 1.00, 95% CI 2-sided [0.97 to 1.04] — [estimate comment as in outcome 1, analysis 1]
Statistical Analysis 2: Comparison: Intervention (Immediate Results) vs Control (Delayed Results); [analysis description as in outcome 1, analysis 2]; Test type: Superiority; Risk Ratio (RR) = 0.91, 95% CI 2-sided [0.74 to 1.12] — [estimate comment as in outcome 4, analysis 2]

9. Secondary Outcome: Count of Participants With SARS-CoV-2 Seroconversion Over 8 Weeks
Description: This outcome will be assessed by comparing SARS-CoV-2 serostatus at baseline (September 2020) and endline (November 2020). Those who were antibody negative at baseline but antibody positive at endline will be considered seroconverters in this study.
Time Frame: Approximately 8 weeks from baseline antibody test.
Measure: Count of Participants; unit: Participants
Arm/Group | Intervention (Immediate Results) | Control (Delayed Results)
Number analyzed (Participants) | 406 | 402
Participants
  Yes | 20 | 22
  No | 386 | 380
Statistical Analysis 1: Comparison: Intervention (Immediate Results) vs Control (Delayed Results); This analysis includes only those participants with a negative antibody test result at baseline to test the association between the treatment condition (immediate vs. delayed test results) and seroconversion. The reference group for this analysis was the control (delayed results) group; Test type: Superiority; Risk Ratio (RR) = 0.94, 95% CI 2-sided [0.52 to 1.71] — This analysis compares the probability of seroconverting during the study period. The reference group for this analysis was the control (delayed results) group

ADVERSE EVENTS:
Time Frame: Eight weeks, from baseline antibody testing to endline antibody testing
Arm/Group | Intervention (Immediate Results) | Control (Delayed Results)
All-Cause Mortality (participants affected / at risk) | 0/536 | 0/540
Serious Adverse Events (participants affected / at risk) | 0/536 | 0/540
Other Adverse Events (participants affected / at risk) | 0/536 | 0/540

LIMITATIONS AND CAVEATS:
As results were disseminated by email, we cannot confirm that everyone in each treatment condition received their results on the expected schedule, or at all. However, operational and survey data we collected indicated that participants received their test results at similar rates in both arms, alleviating concerns of differential intervention uptake.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT04620798/Prot_SAP_000.pdf
  • Informed Consent Form (2020-09-01): https://cdn.clinicaltrials.gov/large-docs/98/NCT04620798/ICF_001.pdf